CLINICAL TRIAL: NCT03168087
Title: The Effect of a Plasmalyte-148 Solution on Blood Coagulation: In Vitro, Volunteer Study Using Rotational Thromboelastometry
Brief Title: Plasmalyte-148 Solution and Blood Coagulation
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Jung Shin, Assistant professor, Seoul National University Bundang Hospital
Other Study IDs: B-1705/395-303
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Blood Coagulation Disorder
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 0% dilution: Blood specimen which was diluted with 0% level using a plasmalyte-148 solution
- 20% dilution: Blood specimen which was diluted with 20% level using a plasmalyte-148 solution
  Interventions: Other: Plasmalyte-148
- 40% dilution: Blood specimen which was diluted with 40% level using a plasmalyte-148 solution
  Interventions: Other: Plasmalyte-148
- 60% dilution: Blood specimen which was diluted with 60% level using a plasmalyte-148 solution
  Interventions: Other: Plasmalyte-148

INTERVENTIONS:
Other: Plasmalyte-148 — Venous blood is taken from 12 healthy volunteers and divided into four specimen bottles, which were diluted with different levels (0%, 20%, 40%, and 60%) using a plasmalyte-148 solution.
  Groups: 20% dilution; 40% dilution; 60% dilution

SUMMARY:
Fluids administered intravenously may alter whole blood coagulation. However, little is known about the dose-response relationships of hemodilution in plasmalyte-148 solution. Investigators have therefore performed the present study to measure the effect of a plasmalyte-148 solution on the coagulation pathway according to the hemodilution level using a rotational thromboelastometry (ROTEM®) tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age: 20 to 65 years
* Body weight > 50 kg
* Volunteers who provided informed consent

Exclusion Criteria:

* Hematologic disease
* Anticoagulant medication

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
FIBTEM | During the rotational thromboelastometry analysis/ an average of 1 hour
  Fibrinolytic pathway values of rotational thromboelastometry analysis/ FIBTEM is not an acronym.

SECONDARY OUTCOMES:
INTEM | During the rotational thromboelastometry analysis/ an average of 1 hour
  Intrinsic pathway values of rotational thromboelastometry analysis/ INTEM is not an acronym.
EMTEM | During the rotational thromboelastometry analysis/ an average of 1 hour
  Extrinsic pathway values of rotational thromboelastometry analysis/ EXTEM is not an acronym.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Jung Shin, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No